CLINICAL TRIAL: NCT02650076
Title: A Study to Investigate the Receptor Occupancy of SK-1405 in Healthy, Caucasian, Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanwa Kagaku Kenkyusho Co., Ltd. (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: MO001A
Record Dates: First submitted 2016-01-05; First posted 2016-01-08 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Pruritus
MeSH Terms: conditions — Pruritus

ARMS (1):
- Healthy (Experimental)
  Interventions: Drug: SK-1405

INTERVENTIONS:
Drug: SK-1405

SUMMARY:
The primary objective is to confirm the target receptor occupancy of SK-1405 and to correlate receptor occupancy with SK-1405 dose and plasma concentration.

The secondary objective is to assess the safety and tolerability of SK-1405 in healthy, Caucasian, male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide written informed consent to participate in this study, as confirmed by signing the informed consent document(s).
* Adult Caucasian male aged ≥20 and ≤50 years.
* Body Mass Index (BMI) of ≥ 20 and ≤ 30 kg/m2.
* Height ≤ 190 cm.
* Subject is a non-smoker or has not smoked in the past 6 months.
* Subject is considered to be in good health in the opinion of the investigator.
* Subject's pre-study clinical laboratory findings are within normal range.
* Subject must be willing and able to comply with all protocol requirements.

Exclusion Criteria:

* Use of prohibited medications as described in the study protocol.
* Current known or suspected history of drug/solvent abuse.
* Current known or suspected history of alcohol abuse or currently drinks in excess of 21 units per week.
* Subjects who have consumed caffeine containing products within 24 hours prior to baseline PET-CT.
* Any concurrent medical, surgical, or psychiatric condition that may affect the subject's ability to meet all protocol requirements during the study duration and/or any significant illness in the investigator's opinion in the 4 weeks before screening.
* Participation in any other clinical study with an investigational drug/device within three months prior to the first day of dosing and after enrolment in the current study.
* Subject has a positive result of HIV screen, hepatitis B screen or hepatitis C screen.
* Subject has had a serious adverse reaction or significant hypersensitivity to any drug.
* Subject has donated 500 mL or more of blood within the three months prior to screening.
* History of neurological conditions.
* Participation in a research study or other radiation exposure which in conjunction with this study would result in additional ionisation radiation exposure exceeding 10 mSv within the last year.
* A contraindication for MRI, including but not limited to, MRI-incompatible pacemakers, recent metallic implants, foreign body in the eye, or other indications as assessed by a standard pre-MRI questionnaire, that preclude the subject undergoing MRI scans.
* Subject has claustrophobia.
* Subjects who have consumed Saint John's wort, red wine, Seville oranges, grapefruit or grapefruit juice within 7 days prior to dosing.
* Subject has a partner who is either pregnant or breastfeeding for the duration of the study.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2016-01; Primary Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
The receptor occupancy of SK-1405 as measured by PET-CT imaging with [11C]-carfentanil | up to 4 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hammersmith Medicines Research, London, London, United Kingdom